CLINICAL TRIAL: NCT04317508
Title: Effectiveness of Benzocaine Gelpatch in Reducing Injection Pain in Pediatric Dental Patients:A Randomized Clinical Trial
Brief Title: Using Anesthetic Gel Patches to Reduce Pain of Palatal Injection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dina Youssef Attia (Other)
Responsible Party: Sponsor-Investigator, Dina Youssef Attia, Assistant lecturer, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Benzocaine gel patch
Record Dates: First submitted 2020-03-12; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Anesthesia, Dental
Keywords: benzocaine; Topical; oral patch; pain; dental anesthesia; children
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Split mouth randomized clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: * Administration of local anesthetic will be video recorded.
  * An independent investigator who is blinded to the type of topical applied will evaluate the outcome from the video recordings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Topicale® topical anesthetic gel patch (Benzocaine 18%)
  Interventions: Drug: Topicale GelPatch (Benzocaine 18%)
- control group (Placebo Comparator): Opahl® topical anesthetic gel (Benzocaine 20%)
  Interventions: Drug: Benzocaine oral gel 20%

INTERVENTIONS:
Drug: Topicale GelPatch (Benzocaine 18%) — Intervention group
  Arms: Intervention group
Drug: Benzocaine oral gel 20% — control group
  Arms: control group

SUMMARY:
Local anesthetic administration step is mandatory step for controlling pain before dental procedures. The aim of this study was to compare effectiveness of topical Benzocaine 18% gel patch form and Benzocaine 20% topical gel in reducing pain during injection of local anesthesia in children receiving dental treatment.

DETAILED DESCRIPTION:
A sample of 50 children ranging in age from 6 to 8 years who need a bilateral dental treatment in the same arch participated in this study. They were healthy children rated 3 or 4 according to Frankl behavioral rating scale. They were selected from the clinic of Pediatric Dentistry Department, Faculty of Dentistry, Alexandria University.

A randomized split mouth design was done in which each child received both tested topical anesthetics on each side of the arch. The topical anesthetic gel patch or the topical gel application was randomly used at the first or second visits. Pain or discomfort was evaluated during injection using sound, eye, motor (SEM) scale, and after injection using faces pain scale- revised (FPS-R).

ELIGIBILITY:
Inclusion Criteria:

1. Children ranging in age from 6 to 8 years.
2. Healthy children with no contraindications of use of local anesthetics.
3. Cooperative behavior according to Frankl's scale scores 3 or 4. (appendix I)
4. Patients needing dental interventions on both sides in the same arch that will require palatal or inferior alveolar nerve block injections.

Exclusion Criteria:

1. Uncooperative children or with intellectual or physical disabilities or medical conditions.
2. Children with acute pain or emergency visits.
3. Children with previous negative dental experience.
4. Children receiving premedications or analgesics 48 hours before testing.
5. children/parents not willing to participate.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-13 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Comparing the tolerability of oral topical anesthetic Topicale GelPatch (Benzocaine 18%) and Benzocaine oral gel 20% during injection | 4 months
  The aim was to reduce pain and discomfort during injection of local anesthesia in pediatric dental patients. Pain or discomfort was evaluated during injection using sound, eye, motor (SEM) scale
  Sound, Eye, Motor scale:
  Grade 1: Comfort
  * Sound: No sound
  * Eye: No signs
  * Motor: Relaxed body and hand
  Grade 2: Mild discomfort
  * Sound: Non specific sound
  * Eye: Dilated without tears
  * Motor: Muscular contractions of hand
  Grade 3: Moderate discomfort
  * Sound: Verbal compliant, louder sound
  * Eye: Tears, sudden eye movement
  * Motor: Sudden body and hand movements
  Grade 4: Severe discomfort
  * Sound: Verbal compliant shouting, crying
  * Eye: Crying, tears all over face
  * Motor: Hand movement for defense, Turning the head to opposite side
Comparing the tolerability of oral topical anesthetic Topicale GelPatch (Benzocaine 18%) and Benzocaine oral gel 20% after injection | 4 months
  Pain or discomfort was evaluated after injection using faces pain scale-revised (FPS-R).
  2- Face Pain Scale- Revised: Scoring the chosen face 0, 2, 4, 6, 8, or 10, counting left to right, so "0" = "no pain" and "10" = "very much pain".

CONTACTS AND LOCATIONS:
Overall Officials: Huda M Ibrahim, BSc, Principal Investigator — Alexandria University; Amina Abdelrahman, PhD, Study Director — Alexandria University; Aly Sharaf, PhD, Study Director — Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bagesund M, Tabrizi P. Lidocaine 20% patch vs lidocaine 5% gel for topical anaesthesia of oral mucosa. Int J Paediatr Dent. 2008 Nov;18(6):452-60. doi: 10.1111/j.1365-263X.2007.00910.x. Epub 2008 Mar 12. PMID 18341564
- [Result] Stecker SS, Swift JQ, Hodges JS, Erickson PR. Should a mucoadhesive patch (DentiPatch) be used for gingival anesthesia in children? Anesth Prog. 2002 Winter;49(1):3-8. PMID 12779107